CLINICAL TRIAL: NCT05994794
Title: A Randomized, Single-Blind, Placebo-Controlled Trial for the Role of a Dietary Supplement in Lowering S-Adenosylhomocysteine (SAH) in Healthy Adults With Elevated Plasma SAH and Normal Homocysteine Levels and Identification of Participants With Elevated Plasma SAH in the General Population Using the MethylQ Score
Brief Title: Role of a Dietary Supplement in Lowering SAH in Healthy Adults With Elevated Plasma SAH and Normal Homocysteine Levels
Acronym: SAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S01-21-01-T0023
Record Dates: First submitted 2023-06-28; First posted 2023-08-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Elevated S-adenosylhomocysteine
Keywords: Methylation; Alpha-GPC; Creatine; Ashwagandha
MeSH Terms: interventions — Creatine; Ashwagandha

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alpha-GPC, Creatine and Ashwagandha (Sensoril®) (Experimental): Two servings (12 capsules) of study products will be taken twice per day with meals, one serving in the morning and one serving the afternoon/evening. One serving consists of 6 capsules. The time difference between the two servings must be at least 6 hours.
  One serving:
  * One capsule of Alpha GPC supplement
  * Four capsules of Creatine monohydrate supplement
  * One capsule of Sensoril (ashwagandha) supplement
  Interventions: Dietary Supplement: Alpha-GPC, Creatine and Ashwagandha (Sensoril®)
- Placebo (Placebo Comparator): Participants will consume one serving (6 capsules), twice per day, with meals at least 6 hours apart.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha-GPC, Creatine and Ashwagandha (Sensoril®) — Other Ingredients: Microcrystalline Cellulose, Rice Fiber, Maltodextrin, Silica, Vegetable Stearate
  Arms: Alpha-GPC, Creatine and Ashwagandha (Sensoril®)
Other: Placebo — Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
S-adenosylhomocysteine (SAH) is the end-product of methylation reactions in the body and the precursor to homocysteine. Elevated SAH in the blood is a reflection of the dysregulation of what is known as the S-adenosylmethionine (SAM) cycle and has been associated with poor health outcomes. The SAM cycle is a series of reversible reactions necessary for the regulation of many processes in the body.

The goal of this clinical trial is to assess the ability of a dietary supplement to support healthy plasma SAH levels in individuals with high plasma SAH.

Participants in the study will attend a total of 4 clinic visits and consume study product daily for 12 weeks.

DETAILED DESCRIPTION:
Methionine, a dietary amino acid commonly found in meats, is processed by the body and yields the by-product S-adenosylhomocysteine (SAH), which then undergoes condensation with ATP to produce S-adenosylmethionine (SAM). SAM is the main methyl donor in many of the reactions that occur in the cell. These methyl reactions are well-known epigenetic mechanisms involved in DNA gene expression. When SAM donates its methyl group in a reaction, it becomes SAH which participates in a reversible reaction with homocysteine. Homocysteine is then removed through re-methylation to methionine using folate and vitamin B12. This decrease in homocysteine levels prevents the over-production of SAH, which can disrupt the methyl reactions throughout the body. Dysregulation of this pathway leads to elevated levels of SAH, which have been associated with various disease states. Therefore, an intervention which can lower SAH may ameliorate the outcomes associated with its elevation. This trial will evaluate the efficacy of a dietary supplement to lower SAH in individuals with elevated SAH and normal homocysteine. In addition, this study aims to explore the correlation between the MethylQ score (derived from 3 questionnaires) and measures of SAH level and the SAM:SAH ratio.

The test product contains alpha-GPC, creatine, and ashwagandha. Individually, these ingredients have been shown to improve levels of either SAH or homocysteine in clinical trials.

Participants will be assigned to either the test product or placebo at a 5:3 and consume study product orally for 12 weeks. Assessment measures will include methylation biomarkers, free cortisol index, mood states and MethylQ score in individuals with elevated SAH levels (≥ 20 nmol/L) and normal homocysteine (≤ 13 µmol/L).

The study will include a screening visit followed by a screening period lasting up to 90 days in duration with a remote check-in via phone call occurring between Day -40 and Day -30 (inclusive) for participants screened more than 30 days prior to the baseline visit on (Visit 2). Following the screening period, participants will attend a baseline visit on Day 1, an interim visit on Day 43 ± 3, and an end of study visit on the day after the 12-week (± 3 days) study product use (Day 85 ± 3). The study will include a total of 4 in-person visit days: a screening visit (Visit 1), a baseline visit (Visit 2), an interim visit (Visit 3), and an EOS visit (Visit 4).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults who are 30 to 75 years of age (inclusive).
2. Have a BMI between 18.5 to 34.9 kg/m^2 (inclusive).
3. In good general health (no uncontrolled diseases or conditions) as deemed by the investigator and is able to consume the study product.
4. Have elevated plasma SAH levels of ≥ 20 nmol/L and normal plasma homocysteine levels of ≤ 13 µmol/L at the screening visit (Visit 1).
5. Individuals with childbearing potential must agree to practice an acceptable form of birth control for a certain timeframe prior to the first dose of study product and throughout the study, including:

   1. use for at least 3 months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), or hormone implant (e.g., Norplant System), or intrauterine devices (e.g., Mirena); or
   2. use for at least 1 month prior to the first dose of study product: double-barrier method, non-hormonal intrauterine devices (i.e., copper), or complete abstinence from sexual intercourse that may result in pregnancy; or
   3. vasectomy of partner at least 6 months prior to the first dose of study product.

   Individuals with the potential to impregnate others must agree to use condoms or other acceptable methods to prevent pregnancy throughout the study. Complete abstinence from sexual intercourse that may result in pregnancy is also acceptable.
6. Agree to comply with concomitant treatment restrictions, permitted time frames and/or conditions listed in Study Protocol (No. S01-21-01-T0023) Section 6.5 (Concomitant Treatments).
7. Have maintained stable dietary habits (including supplement intake), exercise habits and lifestyle for the last 3 months prior to screening and agree to maintain dietary and exercise habits and lifestyle throughout the study.
8. Willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Individuals who are lactating, pregnant or planning to become pregnant during the study as confirmed at the baseline visit (Visit 2).
2. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
3. Currently has COVID-19 or tests positive for COVID-19 within 28 days prior to baseline visit.
4. Currently has any post Covid-19 condition(s) as defined by World Health Organization (WHO) (i.e., individuals with a history of a probable or confirmed SARS-CoV-2 infection, usually three months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis).
5. Have a history of heart disease/cardiovascular disease, uncontrolled hypertension (140/90 or greater mmHg), kidney dysfunction or disease (dialysis or renal failure), hepatic impairment or disease, or Type I or Type II diabetes.
6. Have a history of thyroid disease, major affective disorder, psychiatric disorder (e.g., bipolar disorder) that required hospitalization in the prior year, autoimmune diseases (e.g., multiple sclerosis, Parkinson's, systemic lupus erythematosus, rheumatoid arthritis, etc.), or immune disorder (i.e., HIV/AIDS).
7. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g. dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
8. Have an active malignant disease, except basal or squamous cell skin carcinoma or carcinoma in situ of the uterine cervix.
9. Major surgery in 3 months prior to the screening visit (Visit 1) or planned major surgery during the course of the study.
10. History of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program).
11. Receipt or use of test product(s) in another research study within 28 days prior to baseline or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
12. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
To determine the effect of the Test Product (TP) compared to placebo on plasma S-adenosylmethionine (SAM) concentration. | 12 weeks
  Change from baseline in plasma SAM (nmol/L).
To determine the effect of the TP compared to placebo on plasma S-adenosylhomocysteine (SAH) concentration. | 12 weeks
  Change from baseline in plasma SAH (nmol/L).
To determine the effect of the TP compared to placebo on plasma homocysteine concentration. | 12 weeks
  Change from baseline in plasma homocysteine (umol/L).
To determine the effect of the TP compared to placebo on plasma cystathionine concentration. | 12 weeks
  Change from baseline in plasma cystathionine (umol/dL).
To determine the effect of the TP compared to placebo on plasma cysteine concentration. | 12 weeks
  Change from baseline in plasma cysteine (umol/dL).
To determine the effect of the TP compared to placebo on plasma methionine concentration. | 12 weeks
  Change from baseline in plasma methionine (umol/dL).

SECONDARY OUTCOMES:
To determine the effect of the TP compared to placebo on plasma SAM concentration. | 6 weeks
  Change from baseline in plasma SAM (nmol/L).
To determine the effect of the TP compared to placebo on plasma SAH concentration. | 6 weeks
  Change from baseline in plasma SAH (nmol/L).
To determine the effect of the TP compared to placebo on plasma homocysteine concentration. | 6 weeks
  Change from baseline in plasma homocysteine (umol/L).
To determine the effect of the TP compared to placebo on plasma cystathionine concentration. | 6 weeks
  Change from baseline in plasma cystathionine (umol/dL).
To determine the effect of the TP compared to placebo on plasma methionine concentration. | 6 weeks
  Change from baseline in plasma methionine (umol/dL).
To determine the effect of the TP compared to placebo on plasma cysteine concentration. | 6 weeks
  Change from baseline in plasma cysteine (umol/dL).
To determine the effect of the TP compared to placebo on overall mood state. | 12 weeks
  Change from baseline in total mood disturbance assessed by Profile of Mood States (POMS) questionnaire. A higher score indicates a worse outcome.
To determine the effect of the TP compared to placebo on anger-hostility. | 12 weeks
  Change from baseline in anger-hostility subscore from the POMS questionnaire. A higher score indicates a worse outcome.
To determine the effect of the TP compared to placebo on vigor-activity. | 12 weeks
  Change from baseline in vigor-activity subscore from the POMS questionnaire. A higher score indicates a better outcome.
To determine the effect of the TP compared to placebo on confusion-bewilderment. | 12 weeks
  Change from baseline in confusion-bewilderment subscore from the POMS questionnaire. A higher score indicates a worse outcome.
To determine the effect of the TP compared to placebo on depression-dejection. | 12 weeks
  Change from baseline in depression-dejection subscore from the POMS questionnaire. A higher score indicates a worse outcome.
To determine the effect of the TP compared to placebo on tension-anxiety. | 12 weeks
  Change from baseline in tension-anxiety subscore from the POMS questionnaire. A higher score indicates a worse outcome.
To determine the effect of the TP compared to placebo on friendliness. | 12 weeks
  Change from baseline in friendliness subscore from the POMS questionnaire. A higher score indicates a better outcome.
To determine the effect of the TP compared to placebo on fatigue-inertia. | 12 weeks
  Change from baseline in fatigue-interia subscore from the POMS questionnaire. A higher score indicates a worse outcome.
To determine the effect of the TP compared to placebo on free cortisol index. | 12 weeks
  Change from baseline in the ratio of total cortisol/cortisol-binding globulin (CBG).
To determine the effect of the TP compared to placebo on the MethylQ score. | 12 weeks
  Change from baseline in MethylQ score. A score greater than 30 indicates a worse outcome.

OTHER OUTCOMES:
MethylQ score and Plasma SAH Correlation | Screening, Baseline and Week 12
  To determine a correlation between MethylQ score and plasma SAH level at screening, baseline and Week 12.
MethylQ score and SAM/SAH Ratio Correlation | Screening, Baseline and Week 12
  To determine a correlation between MethylQ score and plasma SAH level at screening, baseline and Week 12.
Post-dose change in Plasma SAH and MethylQ score Correlation | 12 weeks
  To determine a correlation between post-dose changes in plasma SAH level with post-dose MethylQ score.
Post-dose change in SAM/SAH Ratio and MethylQ score Correlation | 12 weeks
  To determine a correlation between post-dose changes in SAM/SAH ratio with post-dose MethylQ score.
Heart rate | 12 weeks
  Change from baseline in heart rate (beats per minute).
Blood pressure | 12 weeks
  Change from baseline in blood pressure (mmHg).
Body weight | 12 weeks
  Change from baseline in weight (kg).
Body mass index | 12 weeks
  Change from baseline in body mass index (BMI) (kg/m^2).
Whole Blood Hemoglobulin | 12 weeks
  Change from baseline in fasting whole blood hemoglobulin (g/dL) between TP and placebo.
Whole Blood Hematocrit | 12 weeks
  Change from baseline in fasting whole blood hematocrit (%) between TP and placebo.
Whole Blood White Blood Cells | 12 weeks
  Change from baseline in fasting whole blood white blood cell count (x10^3/uL) between TP and placebo.
Whole Blood Neutrophils | 12 weeks
  Change from baseline in fasting whole blood neutrophil count (cells/uL) between TP and placebo.
Whole Blood Basophils | 12 weeks
  Change from baseline in fasting whole blood basophil count (cells/uL) between TP and placebo.
Whole Blood Eosinophils | 12 weeks
  Change from baseline in fasting whole blood eosinophil count (cells/uL) between TP and placebo.
Whole Blood Monocytes | 12 weeks
  Change from baseline in fasting whole blood monocyte count (cells/uL) between TP and placebo.
Whole Blood Lymphocytes | 12 weeks
  Change from baseline in fasting whole blood lymphocyte count (cells/uL) between TP and placebo.
Whole Blood Red Blood Cell Count | 12 weeks
  Change from baseline in fasting whole blood red blood cell count (x10^6/uL) between TP and placebo.
Whole Blood Red blood cell distribution width | 12 weeks
  Change from baseline in fasting whole blood red blood cell distribution width (%) between TP and placebo.
Whole Blood Mean Corpuscular Volume | 12 weeks
  Change from baseline in fasting whole blood mean corpuscular volume (fL) between TP and placebo.
Whole Blood Mean Corpuscular Hemoglobin | 12 weeks
  Change from baseline in fasting whole blood mean corpuscular hemoglobin (pg) between TP and placebo.
Whole Blood Mean Corpuscular Hemoglobin Concentration (MCHC) | 12 weeks
  Change from baseline in fasting whole blood MCHC (g/dL) between TP and placebo.
Whole Blood Platelet count | 12 weeks
  Change from baseline in fasting whole blood platelet count (x10^3/uL) between TP and placebo.
Whole Blood Mean platelet volume (MPV) | 12 weeks
  Change from baseline in fasting whole blood MPV (fL) between TP and placebo.
Serum Sodium | 12 weeks
  Change from baseline in fasting serum sodium concentration (mmol/L) between TP and placebo.
Serum Potassium | 12 weeks
  Change from baseline in fasting serum potassium concentration (mmol/L) between TP and placebo.
Serum Chloride | 12 weeks
  Change from baseline in fasting serum chloride concentration (mmol/L) between TP and placebo.
Serum Urea | 12 weeks
  Change from baseline in fasting serum urea concentration (mg/dL) between TP and placebo.
Serum Creatinine | 12 weeks
  Change from baseline in fasting serum creatinine concentration (mg/dL) between TP and placebo.
Estimate glomerular filtration rate (eGFR) | 12 weeks
  Change from baseline in eGFR (mL/min/1.73m^2) between TP and placebo.
Serum Total Protein | 12 weeks
  Change from baseline in fasting serum total protein concentration (g/dL) between TP and placebo.
Serum Albumin | 12 weeks
  Change from baseline in fasting serum albumin concentration (g/dL) between TP and placebo.
Serum Globulin | 12 weeks
  Change from baseline in fasting serum globulin concentration (g/dL) between TP and placebo.
Serum Total Bilirubin | 12 weeks
  Change from baseline in fasting serum total bilirubin concentration (mg/dL) between TP and placebo.
Serum Fasting Glucose | 12 weeks
  Change from baseline in fasting serum glucose concentration (mg/dL) between TP and placebo.
Serum Alkaline phosphatase | 12 weeks
  Change from baseline in fasting serum alkaline phosphatase concentration (U/L) between TP and placebo.
Serum Alanine transaminase | 12 weeks
  Change from baseline in fasting serum alanine transaminase concentration (U/L) between TP and placebo.
Serum Aspartate transaminase | 12 weeks
  Change from baseline in fasting serum aspartate transaminase concentration (U/L) between TP and placebo.
Incidence of adverse events | 12 weeks
  To determine number of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bassem F. El-Khodor, PhD, Principal Investigator — Nutrition Innovation Center, Standard Process Inc.
Locations (1):
- Valiance Clinical Research, South Gate, California, United States

REFERENCES:
- [Background] Kennedy BP, Bottiglieri T, Arning E, Ziegler MG, Hansen LA, Masliah E. Elevated S-adenosylhomocysteine in Alzheimer brain: influence on methyltransferases and cognitive function. J Neural Transm (Vienna). 2004 Apr;111(4):547-67. doi: 10.1007/s00702-003-0096-5. Epub 2004 Feb 4. PMID 15057524
- [Background] Xiao Y, Huang W, Zhang J, Peng C, Xia M, Ling W. Increased plasma S-adenosylhomocysteine-accelerated atherosclerosis is associated with epigenetic regulation of endoplasmic reticulum stress in apoE-/- mice. Arterioscler Thromb Vasc Biol. 2015 Jan;35(1):60-70. doi: 10.1161/ATVBAHA.114.303817. Epub 2014 Oct 30. PMID 25359864
- [Background] Lawson BR, Eleftheriadis T, Tardif V, Gonzalez-Quintial R, Baccala R, Kono DH, Theofilopoulos AN. Transmethylation in immunity and autoimmunity. Clin Immunol. 2012 Apr;143(1):8-21. doi: 10.1016/j.clim.2011.10.007. Epub 2011 Dec 24. PMID 22364920
- [Background] Ganguly P, Alam SF. Role of homocysteine in the development of cardiovascular disease. Nutr J. 2015 Jan 10;14:6. doi: 10.1186/1475-2891-14-6. PMID 25577237
- [Background] Moore LD, Le T, Fan G. DNA methylation and its basic function. Neuropsychopharmacology. 2013 Jan;38(1):23-38. doi: 10.1038/npp.2012.112. Epub 2012 Jul 11. PMID 22781841
- [Background] Troen AM, Lutgens E, Smith DE, Rosenberg IH, Selhub J. The atherogenic effect of excess methionine intake. Proc Natl Acad Sci U S A. 2003 Dec 9;100(25):15089-94. doi: 10.1073/pnas.2436385100. Epub 2003 Dec 1. PMID 14657334
- [Background] Olthof MR, Brink EJ, Katan MB, Verhoef P. Choline supplemented as phosphatidylcholine decreases fasting and postmethionine-loading plasma homocysteine concentrations in healthy men. Am J Clin Nutr. 2005 Jul;82(1):111-7. doi: 10.1093/ajcn.82.1.111. PMID 16002808
- [Background] Innis SM, Davidson AG, Melynk S, James SJ. Choline-related supplements improve abnormal plasma methionine-homocysteine metabolites and glutathione status in children with cystic fibrosis. Am J Clin Nutr. 2007 Mar;85(3):702-8. doi: 10.1093/ajcn/85.3.702. PMID 17344490
- [Background] Korzun WJ. Oral creatine supplements lower plasma homocysteine concentrations in humans. Clin Lab Sci. 2004 Spring;17(2):102-6. PMID 15168891
- [Background] Bonilla DA, Moreno Y, Gho C, Petro JL, Odriozola-Martinez A, Kreider RB. Effects of Ashwagandha (Withania somnifera) on Physical Performance: Systematic Review and Bayesian Meta-Analysis. J Funct Morphol Kinesiol. 2021 Feb 11;6(1):20. doi: 10.3390/jfmk6010020. PMID 33670194
- [Derived] Pohl F, Dominique A, Dufour J, Wang J, Lin XL, Sharif B, Wilson M, Gonzalez L, El-Khodor BF. Lowering plasma S-Adenosylhomocysteine (SAH) in healthy adults with elevated SAH and normal homocysteine using nutritional supplementation. Nutr Metab Cardiovasc Dis. 2025 Dec;35(12):104221. doi: 10.1016/j.numecd.2025.104221. Epub 2025 Jul 5. PMID 40883125